CLINICAL TRIAL: NCT00002524
Title: Pilot Study in AIDS-Related Lymphomas
Brief Title: Combination Chemotherapy in Treating Patients With AIDS-Related Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM93-058; P30CA016672 (NIH); MDA-DM-93058 (Other: UT MD Anderson Cancer Center); NCI-T93-0088D; CDR0000078316 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-10-05 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Lymphoma
Keywords: AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; AIDS-related diffuse large cell lymphoma; AIDS-related immunoblastic large cell lymphoma; AIDS-related small noncleaved cell lymphoma; AIDS-related diffuse mixed cell lymphoma; AIDS-related diffuse small cleaved cell lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Bleomycin; Filgrastim; Granulocyte Colony-Stimulating Factor; Cisplatin; Cyclophosphamide; Cytarabine; Doxorubicin; Etoposide; Fluorouracil; Ifosfamide; Leucovorin; Methotrexate; Methylprednisolone; Methylprednisolone Acetate; Methylprednisolone Hemisuccinate; Pentamidine; Prednisone; Trimethoprim, Sulfamethoxazole Drug Combination; Vincristine; Cortodoxone; Zidovudine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Regimen A (Experimental): Regimen A: 5-Drug Combination Chemotherapy followed by Radiotherapy.
  Interventions: Biological: Bleomycin Sulfate; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride (DOX); Drug: Pentamidine; Drug: Prednisone; Drug: Trimethoprim-Sulfamethoxazole; Drug: Vincristine Sulfate; Drug: Zidovudine (AZT); Radiation: Radiation Therapy
- Regimen B (Experimental): Regimen B: 4-Drug Combination Chemotherapy alternating with 3-Drug Combination Chemotherapy followed, as indicated, by Radiotherapy
  Interventions: Biological: Filgrastim; Drug: Cytarabine; Drug: Doxorubicin Hydrochloride (DOX); Drug: Etoposide; Drug: Ifosfamide; Drug: Methotrexate; Drug: Methylprednisolone; Drug: Pentamidine; Drug: Trimethoprim-Sulfamethoxazole; Drug: Zidovudine (AZT); Radiation: Radiation Therapy
- Regimen C (Experimental): Regimen C: 2-Drug Combination Chemotherapy with Drug Modulation followed, as indicated, by Radiotherapy.
  Interventions: Biological: Filgrastim; Drug: Cisplatin; Drug: Fluorouracil; Drug: Leucovorin calcium; Drug: Pentamidine; Drug: Trimethoprim-Sulfamethoxazole; Drug: Zidovudine (AZT); Radiation: Radiation Therapy

INTERVENTIONS:
Biological: Bleomycin Sulfate
  Other Names: Blenoxane; BLM
  Arms: Regimen A
Biological: Filgrastim
  Other Names: G-CSF; Neupogen
  Arms: Regimen B; Regimen C
Drug: Cisplatin
  Other Names: Platinol; Plationol-AQ; CDDP
  Arms: Regimen C
Drug: Cyclophosphamide
  Other Names: Cytoxan; Neosar
  Arms: Regimen A
Drug: Cytarabine
  Other Names: Ara-C; Cytosar; DepoCyt; Cytarabine arabinosine hydrochloride
  Arms: Regimen B
Drug: Doxorubicin Hydrochloride (DOX)
  Other Names: Adriamycin PFS; Adriamycin RDF
  Arms: Regimen A; Regimen B
Drug: Etoposide
  Other Names: VePesid
  Arms: Regimen B
Drug: Fluorouracil
  Other Names: 5-FU; Adrucil; Efudex; 5-Fluorouracil
  Arms: Regimen C
Drug: Ifosfamide
  Other Names: Ifex
  Arms: Regimen B
Drug: Leucovorin calcium
  Other Names: Citrovorum; Wellcovorin
  Arms: Regimen C
Drug: Methotrexate
  Arms: Regimen B
Drug: Methylprednisolone
  Other Names: Depo-Medrol; Medrol; Solu-Medrol
  Arms: Regimen B
Drug: Pentamidine
  Other Names: Pentam-300
Drug: Prednisone
  Arms: Regimen A
Drug: Trimethoprim-Sulfamethoxazole
  Other Names: SMX; Bactrim; Cotrim; Septra; Sulfamethoprim; Sulfatrim; Sulfoxaprim; Trisulfam; Uroplus; Co-trimoxazole; SMX-TMP
Drug: Vincristine Sulfate
  Arms: Regimen A
Drug: Zidovudine (AZT)
  Other Names: Retrovir
Radiation: Radiation Therapy
  Other Names: RT; Radiotherapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating patients with AIDS-related lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Develop an effective chemotherapy regimen with mild immunosuppressive and myelosuppressive properties to treat patients with AIDS-related lymphoma (ARL) who have severe T4 lymphopenia. II. Estimate the CR rate, lymphoma-free survival, and overall survival of non-T4 lymphopenic patients and patients who present with nonbulky Ann Arbor stage I ARL treated with standard regimens of known effectiveness. III. Evaluate the effects on long-term outlook of concurrent antiretroviral therapy, prophylactic antibiosis with trimethoprim/sulfamethoxazole or aerosolized pentamidine, and prn use of granulocyte colony-stimulating factor for severe myelosuppression.

OUTLINE: Patients are assigned to Regimens A, B, and C according to histology and extent of disease and the degree of immunosuppression as follows: Regimen A: Patients with Ann Arbor stage I intermediate grade or immunoblastic lymphoma with measurable nonbulky disease (less than 7 cm), low LDH (less than 686), and no prior opportunistic infection irrespective of T4 count; also those with nonmeasurable stage I extranodal primaries (infiltration of less than 2/3 of an organ site, e.g., stomach, rectum, esophagus, sinus cavity) irrespective of T4 count. Regimen B: All patients (except primary brain lymphoma patients) not assigned to Regimen A who have T4 counts of at least 200 and no history of opportunistic infection; includes all stages of small noncleaved cell lymphoma and bulky stage I and stages II-IV intermediate grade and immunoblastic lymphoma. Regimen C: Patients not assigned to Regimen A or B, i.e., those with T4 counts less than 200 and/or a history of opportunistic infection and those with primary brain lymphoma. The following acronyms are used: ARA-C Cytarabine, NSC-63878 BLEO Bleomycin, NSC-125066 CDDP Cisplatin, NSC-119875 CF Leucovorin calcium, NSC-3590 CTX Cyclophosphamide, NSC-26271 DOX Doxorubicin, NSC-123127 5-FU Fluorouracil, NSC-19893 G-CSF Granulocyte Colony-Stimulating Factor (Amgen), NSC-614629 IFF Ifosfamide, NSC-109723 MePRDL Methylprednisolone succinate Mesna Mercaptoethane sulfonate, NSC-113891 MTX Methotrexate, NSC-740 PRED Prednisone, NSC-10023 VCR Vincristine, NSC-67574 VP-16 Etoposide, NSC-141540 ZDV Zidovudine, NSC-602670 Regimen A: 5-Drug Combination Chemotherapy followed by Radiotherapy. CHOP-BLEO: CTX; DOX; VCR; PRED; BLEO; followed by involved-field irradiation with megavoltage equipment. Regimen B: 4-Drug Combination Chemotherapy alternating with 3-Drug Combination Chemotherapy followed, as indicated, by Radiotherapy. ASHAP: DOX; MePRDL; ARA-C; CDDP; alternating with IMVP-16: IFF/Mesna; MTX/CF; VP-16; followed, in selected patients with initially bulky localized disease, by involved-field irradiation with megavoltage equipment. Regimen C: 2-Drug Combination Chemotherapy with Drug Modulation followed, as indicated, by Radiotherapy. FLEP: 5-FU/CF/CDDP; followed, in selected patients with initially bulky localized disease, by involved-field irradiation with megavoltage equipment. Prior to starting chemotherapy, patients with primary brain lymphoma receive a course of cranial irradiation using accelerator beams with photon energies of 6-15 MV.

PROJECTED ACCRUAL: Up to 92 patients (10 for Regimen A, 28 for Regimen B, 54 for Regimen C) will be entered over 3 years. If there are no CRs among the first 6 patients on Regimens A and B or the first 19 patients on Regimen C, accrual to that regimen will cease. If more than 4 infectious deaths occur among the first 10 patients or if the rate of disease progression exceeds 20% on any regimen, further accrual to that regimen will cease.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Previously untreated, HIV-related intermediate- and high-grade lymphoma with no previous diagnosis of Kaposi's sarcoma Pathology reviewed at M.D. Anderson Cancer Center

PATIENT CHARACTERISTICS: Age: Over 15 Performance status: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: For patients with T4 less than 200 and those with primary brain lymphoma: Creatinine no greater than 2.0 mg/dL (unless entry approved by principal investigator) Other: Serious intercurrent illness must be discussed with the principal investigator Infectious disease consultation required for complex infections Medications for other conditions allowed provided no adverse interaction with protocol therapy occurs No previously diagnosed Kaposi's sarcoma or other malignancy

PRIOR CONCURRENT THERAPY: No prior therapy for lymphoma No concurrent chemotherapy

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 1993-06; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Clinical Response | 3 Years
  Clinical Responses categorized by: Complete Response (CR), Partial Response (PR), Minor Response, Stable Disease or Progressive Disease

CONTACTS AND LOCATIONS:
Overall Officials: Peter W. McLaughlin, MD, Study Chair — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - University of Texas - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org